CLINICAL TRIAL: NCT06110455
Title: Effects of Neuromuscular Training Compared to Progressive Resistance Training on Patients With Anterior Knee Pain. A Randomized Controlled Trial
Brief Title: Neuromuscular Training Compared to Progressive Resistance Training for Patients With Anterior Knee Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Savvas Spanos, Official Title: Head of Human Performance and Rehabilitation Laboratory of the Physiotherapy Department, University of Thessaly
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NMT PRT Thess
Record Dates: First submitted 2023-10-18; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Anterior Knee Pain Syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — Papaverine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuromuscular Exercise Training (NMT) (Experimental): The 8-week exercise intervention program consists of group sessions of Neuromuscular training supervised by a physical therapist 3 times per week. Patients will be taught and familiarized with the proper way to do the exercises on a separate day prior to the start of their actual rehabilitation program.
  Each session consists of a 5 minute submaximal warm-up followed by 25 minutes of NMT.
  Every 2 weeks, there will be a progression that will be achieved by increasing the difficulty level of each exercise. We will take under consideration the individuality each patient has on how much progression is needed every two weeks and it will be done by maintaining a proper quality of performance, minimal exertion and control of the movement. Participants will be given special equipment including sliders and elastic tubing
  Interventions: Other: Neuromuscular Training exercises
- Progressive Resistance Training (PRT) (Experimental): The 8-week exercise intervention program consists of group sessions of progressive resistance training supervised by a physical therapist 3 times per week. Patients will be taught and familiarized with the proper way to do the exercises on a separate day prior to the start of their actual rehabilitation program.
  Each session consists of a 5 minute submaximal warm-up followed by 25 minutes of PRT, targeting hip and knee muscles, such as hip abductors, knee flexors and extensors. The exercise intensity will be monitored by the physical therapist, as determined by the patients' ability to complete 3 sets of 8-12 repetitions for a given exercise and a Borg Rating of Perceived Exertion (RPE) of 6-8.
  Every 2 weeks, progression will be achieved by changing the resistance based on VAS and RPE, with an elastic tubing
  Interventions: Other: Hip and Knee Muscular Strength exercises

INTERVENTIONS:
Other: Neuromuscular Training exercises — The 8 week exercise intervention consists of 25 minute group sessions of Neuromuscular training supervised by a physical therapist.
  Arms: Neuromuscular Exercise Training (NMT)
Other: Hip and Knee Muscular Strength exercises — The 8 week exercise intervention consists of 25 minute group sessions of progressive resistance training, supervised by a physical therapist.
  Arms: Progressive Resistance Training (PRT)

SUMMARY:
The primary aim of this randomized control trial is to investigate patients' with anterior knee pain if a neuromuscular training program (NMT) has better results in pain and functionality, than an ordinary progressive resistance training program (PRT). Pain will be measured via a visual analog scale for pain (VAS) and functionality via questionnaires such as Kujala and the Greek version of the Modified Baecke Questionnaire (mBQ) and functional tests such as the Anterior Lunge test, Step up/down, squat, balance and reach test. The secondary aims are to investigate the:

1. Hip and knee muscles strength, which will be measured with the Kinvent K-Push dynamometer. Strength will be measured before and after the rehabilitation programs (at baseline and after 8 weeks of intervention).
2. Balance, will also be measured to see the effects of the NMT program.
3. Kinesiophobia, which will be measured with the Tampa Scale
4. Dynamic Knee Valgus, via the Single Leg Landing and Single Leg Squat tests

DETAILED DESCRIPTION:
Participants will be randomized into two groups: PRT or NMT. All sessions will be conducted in group sessions, with one physical therapist/researcher supervising the exercises. Patients will be taught on how to correctly do the exercises beforehand from trained physical therapists. Outcomes will be measured in person at baseline and after 8 weeks of treatment, the exercises will be supervised remotely. The duration of the intervention program will be 8 weeks, with 3 sessions per week with at least one day resting in between, totaling 24 training sessions.

The NMT intervention sessions consist of a 5 minute submaximal warm-up, followed by 25 minutes of NMT with exercises focused on functional and core stability, strength, agility, proprioception, balance, landing, plyometrics and coordination. The training sessions will consist of 5 different exercises. Each of them will be performed for 2 sets, and depending on the exercise either for 8 to 10 reps or for 30 seconds. In between the sets and the exercises there will be a 30 sec rest period. The exercises will be focused on the lower limb which has anterior knee pain and on the core. Four levels of difficulty will be given for each exercise to allow progression. Progression will be individualized for each patient. Every 2 weeks, there will be a progression that will be achieved by changing the exercise gradually, making it harder, or/and changing the support surface.

The PRT intervention will also consist of a 5 minute submaximal warm-up, followed by 25 minutes of the PRT exercises, targeting the hip and knee muscles. The program will consist of 5 different exercises, which each of them will focus on a different muscle group (hip abductors, knee extensors and knee flexors). Each exercise will be performed in sets of 3 of 10 repetitions and there will be a 30 sec rest period between sets and exercises.

Progression will be done by increasing the resistance and by increasing the range of motion. The exercise intensity will be monitored by the researcher, as determined by the patient's ability to complete 3 sets of 8-12 repetitions for a given exercise and a Borg Rating of Perceived Exertion (RPE) of 6-10. The progression will be done safely, based on VAS, patients tolerance and movement quality.

Adherence to the program for both groups will be assessed by the total number of training sessions performed in 8 weeks (total=24 training sessions).

ELIGIBILITY:
Inclusion Criteria:

* Pain ≥ 3 months
* Pain VAS now ≥ 3
* 18-40 y/o
* No pain relief medicine 2 weeks prior to the program
* Kujala 50-80
* Pain during squat, knee bending, palpation, isometric contraction on 60°, long sitting, jumping, step up/down, running.
* Theatre sign
* Positive functional tests: grind test, 45 sec anterior knee provocation, McConnel

Exclusion Criteria:

* Patellar dislocation
* Lower extremity surgery
* Ligament instability
* Rheumatoid Arthritis
* Osteoarthritis
* Tendinopathy
* Meniscus tear
* Ligamentous knee injury or laxity
* Bursitis
* Sinding Larsen Johansson Syndrome
* Previous pathology
* Low back surgery
* Metabolic diseases
* NSAIDs for extended period of time
* Cardiorespiratory diseases
* Sacroiliac joint pain
* Pregnancy
* Physical therapy 2 months ago

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2023-02-02 (Actual); Primary Completion 2023-12-15 (Estimated); Study Completion 2024-05-15 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | Measured at baseline and at the end of the program (week 8)
  Pain will be assessed by a numeric Visual Analogue Scale (VAS), where patients will be asked how much their pain level is. Maximum Score Will be a 10, which is the worst pain they ever felt and minimum score will be 0, which is no pain. Higher scores indicate more pain.
Functionality | Measured at baseline and at the end of the program (week 8)
  Functionality will be assessed by the greek translated version of the Kujala Questionnaire, which is dedicated to assess the functionality of patients with Anterior Knee Pain. The questionnaire is consisted of 13 questions, the maximum score is 100 and minimum score is 0. The lower the score, the less functional the person is.

SECONDARY OUTCOMES:
Stability/Balance | Measured at baseline and at the end of the program (week 8)
  Stability and balance will be assessed via the Y-balance test as well
Strength | Measured at baseline and at the end of the program (week 8)
  Muscle strength of hip and knee muscles will be assessed with the Hogan hand-held dynamometer
Kinesiophobia | Measured at baseline and at the end of the program (week 8)
  Kinesiophobia will be assessed with The Tampa Scale of Kinesiophobia (TSK). It is consisted of 17 items and minimum score is 17 and maximum score is 68. Higher scores indicate an increased level of Kinesiophobia.
Dynamic Knee Valgus | Measured at baseline and at the end of the program (week 8)
  It will be assessed via the Single Leg Landing and Single Leg Squat tests and we will calculate the angle using the Kinovea application

CONTACTS AND LOCATIONS:
Locations (1):
- University of Thessaly, Lamia, Central Greece, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hott A, Brox JI, Pripp AH, Juel NG, Paulsen G, Liavaag S. Effectiveness of Isolated Hip Exercise, Knee Exercise, or Free Physical Activity for Patellofemoral Pain: A Randomized Controlled Trial. Am J Sports Med. 2019 May;47(6):1312-1322. doi: 10.1177/0363546519830644. Epub 2019 Apr 8. PMID 30958707
- [Background] Willy RW, Hoglund LT, Barton CJ, Bolgla LA, Scalzitti DA, Logerstedt DS, Lynch AD, Snyder-Mackler L, McDonough CM. Patellofemoral Pain. J Orthop Sports Phys Ther. 2019 Sep;49(9):CPG1-CPG95. doi: 10.2519/jospt.2019.0302. PMID 31475628
- [Result] Bennell KL, Egerton T, Wrigley TV, Hodges PW, Hunt M, Roos EM, Kyriakides M, Metcalf B, Forbes A, Ageberg E, Hinman RS. Comparison of neuromuscular and quadriceps strengthening exercise in the treatment of varus malaligned knees with medial knee osteoarthritis: a randomised controlled trial protocol. BMC Musculoskelet Disord. 2011 Dec 5;12:276. doi: 10.1186/1471-2474-12-276. PMID 22141334